CLINICAL TRIAL: NCT02387190
Title: Effectiveness of Telenursing Program on Lung Function of Heart Failure Patients: a Randomized Clinical Trial Protocol
Brief Title: REmoTe TelenURsiNg on Lung Function of Heart Failure Outpatients
Acronym: RETURN-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Bahia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado da Bahia (Other)
Responsible Party: Principal Investigator, Carolina de Souza-Machado, NP, PhD, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RETURN-001; RETURN-001 (Other Grant/Funding Number: FAPESB - 8157/2013)
Record Dates: First submitted 2014-05-14; First posted 2015-03-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Lung function test; Telenursing; Morbidity; Mortality; Quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telenursing monitoring (Experimental): The protocol for telenursing allows the realization of standardized professional contacts with the patient and educational approach It is possible through questions and answers coded, that indicate the need for educational intervention or reinforcement of appropriate health behavior.1) Contact the patient by telephone, weekly; 2) Distribution and explanation of the educational booklet; 3) Filling a diary of symptoms and signs; 4) Record, management and markdown visits in case of non-elective visits, hospitalization or fatal episodes. Also, the following aspects shall be observed: help requests associated with illness, adaptations for living with the disease, effects of drugs in daily life, availability of financial resources for disease management, self-image; emotional and social support.
  Interventions: Other: Telenursing monitoring
- Control group (No Intervention): Placebo is considered as standardized education

INTERVENTIONS:
Other: Telenursing monitoring — The telenursing program protocol is based on:
  1. Contact the patient by telephone, weekly;
  2. Distribution and explanation of the educational booklet;
  3. Filling a diary of symptoms and signs; 4) Record, management and markdown visits in case of non-elective visits, hospitalization or fatal episodes. Also, the following aspects shall be observed: help requests associated with illness, adaptations for living with the disease, effects of drugs in daily life, availability of financial resources for disease management, self-image; emotional and social support.
  Arms: Telenursing monitoring

SUMMARY:
Pulmonary dysfunction presented in patients with heart failure is observed as a decrease of maximal aerobic capacity compared to healthy people. Lung function deterioration manifests, in the presence of muscle fatigue and dyspnea on exertion, loss of functional capacity, and activities limitation of daily living. Those manifestation influence the perception of quality of life of patients1.

Patients with heart failure need to develop changes in lifestyle and daily activities aiming to maintain clinical control and prevent the onset of complications and disabilities. If these changes are not often performed, they might carry bigger burden to for the individual and their family and for the healthcare system due to increasing of morbidity and mortality between those patients2.

Systematic reviews conducted in developed countries (USA3, UK4 and Canada5) and developing countries (Colombia6) have shown that telehealth can produce positive effects in individuals with chronic diseases as heart failure. This kind of intervention seems to be effective in preventing hospitalizations and non-elective emergency visits.

In Brazil, telenursing is still a non-standardized and non-diffused intervention. In this perspective, telenursing represents soft new tools to provide quality care. It certainly allows the orientation and training of patients, the permanence of them at home, reduces unnecessary hospitalization. Additionally, this intervention, allows the management of nursing time and strengthens their professional autonomy7.

The principal aim of this study is to describe the protocol to be used in MRE study. The objective of MRE trial is to test the hypothesis that telenursing contributes to the improvement in lung function over the medium term, in patients with heart failure under continuous education.

DETAILED DESCRIPTION:
METHODS STUDY DESIGN It will be a blinded- controlled-randomized clinical trial in parallel-group, with six months follow-up. The trial protocol will be performed in referral outpatient center that accompany patients with heart failure. This unit is part of the public health system in the city of Salvador - Bahia, the second largest city in Northeast of Brazil. The Brazilian health system is one of the largest public health systems in the world. Ensures full access, universal and free to the entire population of the country. Bolstered by a broader concept of health, the health system was created in 1988 by the Brazilian Federal Constitution, to be the health system of more than 180 million Brazilians.

Run-in

The run-in period will last 15 days. After the run-in, eligible patients will be part of the study, according the following criteria:

1. To participate in a telenursing education program;
2. To fill-in a diary of symptoms and signs, daily;
3. To receive calls from the research team weekly;
4. To have attendance at appointment between window of 15 days before or after the scheduled date;
5. To be predisposed to performing spirometry testing, six-minute walk test, pulse oximetry, electrocardiography, and to respond questionnaires about quality of life and scales of dyspnoea.

Wash out

After beginning the project, patients who present the following criteria must be excluded:

1. Pregnancy;
2. Hospitalization for more than 30 days;
3. Do not attend monthly visit inside the search window of 15 days before or after the scheduled date;
4. To change of residence address among states that preclude attendance at scheduled visits;
5. Death;
6. To discharge outpatient clinic of the Hospital of study;
7. Subsequent diagnostic of acute or chronic respiratory disease or other physical/mental condition that makes it impossible to participate in the study;
8. To Cease to participate in telenursingprogram or that study.

RANDOMIZATION

The sample size calculation was performed in Sealed Envelope TM program. 156 patients will be needed (78 per group), using the following indicators: confidence level 95%, 5% maximum error permitted, statistical power of 90% for detecting elevation of the primary endpoint by 12% in the experimental group. After applying the inclusion and exclusion criteria, two groups will be sourced from the randomization and will be allocated into case group and control group without replacement. All subjects included will be assigned a three-digit sequential number (eg. 000-999). These numbers will be fed into groups of four patients with similar characteristics. After that, blok size randomization will be procedure in specific software (www.randomization.com).

INTERVENTIONS The control group will receive standard treatment and monitoring for heart failure from the ambulatory staff where the study will be performed, including pharmacotherapy and health education, as recommended by the health team. The intervention group will receive the standard treatment and ongoing follow-up as well as monitoring by telenursing for a period of 6 months (24 weeks).

The application of remote nursing monitoring program shall establish contact with the participants for six months, through weekly telephone contacts on days and times to be accorded between them. We expected duration of 5 to 10 minutes per call. The team that performs the intervention will explain the content of foreseen contacts with educational approach, allowing the participant a moment to comment and clarification of final questions.

After conclusion of the study, the control group also will receive telenursing intervention if it is proven benefits through this study. The protocol for telenursing intervention deployed can continue in the specialized outpatient clinic and other chronic diseases programs, if proven their benefit.

Implementation of the Program of Telenursing The program of telenursing will consist in weekly contact with patients with heart failure with functional class I, II and III. For the development of telenursing, it will be distributed to the study staff a protocol for remote monitoring practices in nursing and a form of individualized remote monitoring (appendix A and B). Intervention group will be receive educational and support materials (educational booklet and diary of signs and symptoms).

The protocol for telenursing allows the realization of standardized professional contacts with the patient and educational approach It is possible through questions and answers coded, that indicate the need for educational intervention or reinforcement of appropriate health behavior.

The telenursing program protocol is based on: 1) Contact the patient by telephone, weekly; 2) Distribution and explanation of the educational booklet; 3) Filling a diary of symptoms and signs; 4) Record, management and markdown visits in case of non-elective visits, hospitalization or fatal episodes. Also, the following aspects shall be observed: help requests associated with illness, adaptations for living with the disease, effects of drugs in daily life, availability of financial resources for disease management, self-image; emotional and social support.

The protocol is individualized according to the needs identified in the monthly consultation and/or weekly contact for telenursing calls. The protocol addresses the themes: information of health education about the pathology; monitoring the signs and symptoms; adherence to treatment; healthy eating and weight control; breathing exercises; cardiovascular and pulmonary risk factors; physical, occupational and sexual activity; emotional and social support. It functions as a guiding instrument for telenursing, and it is useful in the clinical management of diseases, improvement of self-care, strengthening communication and humanization in relations between professionals and users of health services.

These items will be addressed in alternate calls to avoid wear and loss of information over the phone. Before finalizing the calls, will be offered the individual a moment to express doubts or make other settings regarding the intervention. The nurse is expected to write a report at the end of the calls, by checking the form of individual remote monitoring. All calls will be recorded through Skype and MP3 Skype Recorder software.

The educational booklet containing information about the heart failure and a diary of symptoms and signs will be distributed to the participants, being nurse attribution explain it to them. The booklet developed is a support material for conducting health education by telenursing, illustrated, aimed at answer typical questions, easy to handle and transport, simple visual communication, including to be accessible to individuals with limited understanding of written language. It is a suitable material for the use of the individual as well as the assistance of parents, family members, caregivers and other health professionals and students.

Moreover, after the first contact, will be developed an intervention plan for each individual, according to the needs identified after analysis of medical records and for the nursing consultation. The plan may be modified according to the needs that are identified through the telenursing calls.

Procedures BASELINE: First a baseline period will be held in which, for all individuals enrolled in the study. Following questionnaires will be applied: sociodemographic and clinical characterization formulary; quality of life (Minnesota Living with Heart Failure Questionnaire - MLHFQ); Baseline Dyspnoea Index by Mahler; and electrocardiogram will be performed. When all participants pass through the baseline period, will be preceded randomization and implementation of Visit 01.

Also in this period, a pilot of the telenursing will be made, in which seven study participants will undergo intervention in order to identify necessary changes and adjustments.

VISIT 01 (start of run-in):

For both groups: Application of structured interviews for data collection of socio-demographic and clinical characterization formulary; Application of quality of life questionnaire (MLHFQ); The questionnaire of Baseline Dyspnea Index by Mahler; Conducting pulmonary function test spirometry by a technician certified by the Brazilian Society of Pulmonology; Achievement Test six-minute walk; Measurement of clinical data (pulse oximetry, electrocardiogram, measurement of anthropometric data).

Intervention group: will be explained and distributed a educational booklet and a journal of signs and symptoms. Remote monitoring procedures with nursing continuing education will be explained, collecting best times of contact, collecting phones (personal, neighbors, to run errands, pay phone in the street of residence and mobile phone). On this same visit individuals will be informed of the weekly telephone monitoring and monthly outpatients seen for six months.

Will be provided a standardized health Education for the control group and the intervention group.

VISIT 02, 03, 04, 05:

For both groups: in the days of their regular attendance in the ambulatory will be held: standardized education; reviewed medical clinic (the regular ambulatory); the questionnaires and scales (MLHFQ and Baseline Dyspnoea Index Mahler).

Intervention group: The sessions once a month will be held during the six months of data collection. There will be continuity of telenursing directed to continuing education, weekly.

VISIT 06: all related procedures will be carried out in other visits and additionally walk test six minutes, spirometry, electrocardiogram and pulse oximetry.

ASSESSMENT

1. Sphygmomanometer - Brand: Missouri.
2. Electrocardiograph - Brand: EMAI - Model: 3-channel, 12 simultaneous leads, Graphic Display: LCD 12.8 x 6.4 cm, 12 Outlets EX03.
3. Portable Spirometer for Lung Function Assessment, Brand: KOKO MOE FERRARIS USB.
4. Stethoscope - Brand: Missouri
5. Pulse Oximeter - Brand: Oxilife, Model: Plus Cmos Drake
6. Notebook, Intel Core i5-3210M processor 2.5 GHz, 6GB Memory, 750GB HD, 14-inch LED screen.
7. Headphone - Brand: Trust Model: Quasar 16904.

STATISTICAL ANALYSIS PLAN Descriptive statistics will be used to characterize the individuals search. The analysis of continuous variables will be through measures of central tendency and dispersion; categorical variables will be analyzed using proportions. The difference between proportions will be calculated using the chi-square test. Association tests will be performed. For correlations, the Pearson or Spearman tests depending on the normality of information or number of empty cells are proceeded. Additionally, the risk factors are analyzed according to the cutoff score of quality of life. We will use multivariate linear regression to verify association between risk factors and QoL. FIT equations will be done. There will be also analysis by protocol and by intention to treat. Analyzes stratified by age also compose the statistical plan. The information collected will be fed into a database and analyzed using SPSS 20.0 software (Statistical Package for Social Sciences). Statistically significant values with an interval of confidence greater than or equal to 95% will be considered.

ELIGIBILITY:
Inclusion Criteria:

1. With prior medical diagnosis of heart failure with functional class I, II or III, in accordance to New York Heart Association (NYRA)8.
2. In regular follow-up for at least six months at the study site. Regular follow will be considered when in the period of six months the individual attend at least 2/3 of the scheduled appointments of outpatient unit and 100% of run-in period appointments.
3. With dyspnoea or spirometric volumes evidencing deterioration of lung function.
4. With cognitive conditions to be interviewed.
5. With no medical restrictions to perform spirometry testing and six-minute walk test.
6. With clinical control of the heart failure.

Exclusion Criteria:

1. With psychiatric disorders;
2. Who do not meet eligibility criteria after run-in period;
3. With severe acute or chronic pulmonary disease;
4. Who change clinical parameters during the data collection (severe dyspnoea, peripherical oxygen saturation below 95%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Lung function volumes | Expected average of 6 months
  Evaluation will be done in the V6 compared to V1, only. Baseline has no spirometry test

SECONDARY OUTCOMES:
Related quality of life | Expected average of 6 months
  Minnesota living with heart failure questionnaire
Functional capacity | Expected average of 6 months
  Functional capacity will be evaluated using Six-minutes walking test. Visits are done monthly (avarage)
Morbidity | Weekly during telenursing monitoring (Expected average of 6 months)
  Telenursing monitoring occurs every week during six months in the intervention group (24 weeks)
Mortality | Weekly durng telenursing monitoring program (Expected average of 6 months)
  Telenursing monitoring occurs every week during six months in the intervention group (24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Souza-Machado, PhD, Study Chair — Federal University of Bahia; Carolina Santos, NP, Principal Investigator — Federal University of Bahia; Bárbara Sueli Moreira, NP, Principal Investigator — Federal University of Bahia; Loyane Stenzel, NP, Principal Investigator — Federal University of Bahia
Locations (1):
- Ana nery Hospital, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Rodriguez-Gazquez Mde L, Arredondo-Holguin E, Herrera-Cortes R. Effectiveness of an educational program in nursing in the self-care of patients with heart failure: randomized controlled trial. Rev Lat Am Enfermagem. 2012 Mar-Apr;20(2):296-306. doi: 10.1590/s0104-11692012000200012. English, Portuguese, Spanish. PMID 22699730
- [Background] Riley JP, Gabe JP, Cowie MR. Does telemonitoring in heart failure empower patients for self-care? A qualitative study. J Clin Nurs. 2013 Sep;22(17-18):2444-55. doi: 10.1111/j.1365-2702.2012.04294.x. Epub 2012 Nov 27. PMID 23185992